CLINICAL TRIAL: NCT03691532
Title: Postprandial Fat Metabolism Following an Acute Exercise Bout in Persons With Spinal Cord Injuries
Brief Title: Postprandial Lipid Tracer and Exercise in Spinal Cord Injury
Acronym: PPLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Kevin Allen Jacobs, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20180450
Record Dates: First submitted 2018-06-25; First posted 2018-10-01 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Spinal Cord Injuries
Keywords: lipemia; feeding; paraplegia; tetraplegia; physical activity; macronutrient metabolism
MeSH Terms: conditions — Spinal Cord Injuries; Hyperlipidemias; Paraplegia; Quadriplegia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Mixed-crossover: three separate groups (paraplegia, tetraplegia, and neurologically intact) undergo two conditions (seated control and exercise) in a randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Seated control (CON) (Experimental): Participants remain seated in their habitual wheel chair for ~60 min (duration of exercise performed in other arm). Following the intervention they are fed a liquid meal.
  Interventions: Behavioral: Seated control (CON); Behavioral: Liquid meal
- Arm cycle exercise (ACE) (Experimental): Participants complete continuous arm cycle exercise (ACE) for ~60 min. Following the intervention they are fed a liquid meal.
  Interventions: Behavioral: Arm cycle exercise (ACE); Behavioral: Liquid meal

INTERVENTIONS:
Behavioral: Seated control (CON) — Seated rest
  Arms: Seated control (CON)
Behavioral: Arm cycle exercise (ACE) — Arm cycling at a continuous power output
  Arms: Arm cycle exercise (ACE)
Behavioral: Liquid meal — Liquid meal of 0.5 L volume containing 20 kcal/kg fat free mass (FFM) and 5 mg/kg FFM of uniformly 13-carbon labeled palmitate ([U-13C]palmitate) at a macronutrient distribution of 50% carbohydrate, 35% fat, and 15% protein (by kcal).

SUMMARY:
This study investigates the effect of upper extremity exercise on postprandial lipemia (PPL) in persons with spinal cord injury (SCI). Participants are measured at rest and fed a standardized meal following seated rest (CON) or arm cycling exercise (ACE). The meal is infused with "stable isotope lipid tracers" that allow for determination of the end fates of the fat in the meal.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) results in dysregulation of fat metabolism that increases the risk of morbidity and mortality from cardioendocrine disease. Excessive accumulation of visceral fat after SCI is a serious risk component for cardioendocrine disease and results in part from pronounced hypertriglyceridemia following ingestion of fat-containing meals (i.e., exaggerated postprandial lipemia; PPL). Although exaggerated PPL is well documented in persons with SCI, its etiology is unknown. Specifically, it remains to be determined to what extent exaggerated PPL in those with SCI results from impairments in the use of exogenous (dietary) and/or endogenous (stored) fats. Additionally, it is not known if exercise improves postprandial fat use in a manner that alleviates the exaggerated PPL in this population and reduces the risk of cardioendocrine disease.

The objective of the this study is to examine the mechanisms of exaggerated PPL in those with SCI and the effects of an acute pre-meal exercise bout by employing novel stable isotope tracer techniques. In persons without SCI, it is well established that pre-meal exercise lowers PPL in part by improving the use of exogenous and endogenous fats. While muscle atrophy and blunted sublesional sympathetic activity following SCI may hinder fat use, preliminary data indicate that fat use is increased during recovery from exercise in the postabsorptive (fasted) state in this population. Thus, the investigators hypothesize that decreased use of exogenous and endogenous fats contributes to exaggerated PPL in SCI, and that pre-meal exercise will reduce PPL due to increased use of both fat sources.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-60 years.
* For the spinal cord injury subgroups, the participant's injury will be:

  * neurologically stable,
  * American Spinal Injury Association (ASIA) Impairment Scale A-C,
  * and will have occurred > 1 year from the testing date.

Exclusion Criteria:

* Existing diagnosis of cardiovascular disease or diabetes.
* Contraindication to exercise (ACSM Guideline, 10th edition).
* Lower extremity fracture or dislocation within 6 months of participation.
* History of head injury or seizures.
* Inability to consent.
* Restrictions in upper extremity range of motion that would prevent an individual from achieving an unhindered arm cycling motion or moving throughout a range needed to perform resistance maneuvers.
* A pressure ulcer at ischial/gluteus, trochanteric, sacral, or heel sites within the last 3 months.
* Imprisonment in state or federal jail or prison.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Rates of postprandial exogenous vs. endogenous fat use | 400 minutes
  Indirect calorimetry data (rates of CO2 production and O2 consumption) will be input into stoichiometric equations to calculate the rate of whole body fat oxidation (grams/minute). Breath carbon-13 carbon dioxide (13CO2) enrichment data combined with the rate CO2 production from indirect calorimetry will allow for the determination of the individual rates of exogenous and endogenous fat use.

SECONDARY OUTCOMES:
Contribution of exogenous fat to postprandial changes in plasma triglycerides | 400 minutes
  Carbon-13 palmitate ([U-13C] enrichment data will allow for the determination of the contribution of exogenous fat to the total blood triglyceride concentration. The contribution of endogenous fat to the total blood triglyceride concentration will be calculated by subtracting the exogenous fat contribution from the total blood triglyceride concentration.
Concentration of fats in the blood | 460 minutes
  Concentration of triglycerides, non-esterified fatty acids, and glycerol in the blood before and after a test meal.
Concentration of sugar in the blood | 460 minutes
  Concentration of glucose in the blood before and after a test meal.
Concentration of hormones in the blood | 460 minutes
  Concentration of insulin and catecholamines in the blood before and after a test meal.
Markers of systemic inflammation | Baseline
  Concentration of high-sensitivity C-reactive protein (hs-CRP) in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Jacobs, PhD, Principal Investigator — University of Miami
Locations (1):
- Lois Pope Life Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No